CLINICAL TRIAL: NCT00028093
Title: Combination of Pegylated Interferon and Ribavirin as Therapy for Patients With Chronic Hepatitis C With and Without Renal Disease
Brief Title: Pegylated Interferon and Ribavirin to Treat Chronic Hepatitis C With and Without Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yaron Rotman, M.D., Asst. Clinical Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020065; 02-DK-0065 (Other: NIH Clinical Center)
Record Dates: First submitted 2001-12-11; First posted 2001-12-12 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis; Cirrhosis; Hepatitis C Virus; Hemolysis; Ribavirin; Alpha Interferon; Peginterferon; Antiviral Agents; Viral Hepatitis; Hemolytic Anemia; Renal Failure; Renal Dialysis; Hepatitis; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis, Chronic; Fibrosis; Hepatitis C; Hemolysis; Anemia, Hemolytic; Renal Insufficiency; Hepatitis | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pefinterferon+Ribavirin (Experimental): Patients with chronic hepatitis C virus (HCV) infection genotype 1 peginterferon alpha-2a, 180 ug subcutaneous once weekly and weight-based oral ribavirin (1000 mg daily for patients <75 kg and 1200 mg daily for patients >=75 kg) for 48 weeks
  Interventions: Drug: Peginterferon alfa-2a with Ribavirin
- Peginterferon (Active Comparator): patients with chronic hepatitis C virus (HCV) infection genotype 1 were given peginterferon-alpha-2a, 180 ug subcutaneous once weekly for the first 4 weeks of therapy, after which peginterferon was continued at the same dose and weight-based oral ribavirin was added and continued for an additional 44 weeks.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a with Ribavirin — Eligible patients were given peginterferon alpha-2a, 180 ug subcutaneous once weekly and weight-based oral ribavirin (1000 mg daily for patients <75 kg and 1200 mg daily for patients >=75 kg) for 48 weeks
  Arms: Pefinterferon+Ribavirin
Drug: Peginterferon alfa-2a — Eligible patients were given peginterferon-alpha-2a, 180 ug subcutaneous once weekly for the first 4 weeks of therapy, after which peginterferon was continued at the same dose and weight-based oral ribavirin was added and continued for an additional 44 weeks.
  Arms: Peginterferon

SUMMARY:
This study will examine the effectiveness of pegylated interferon, or peginterferon (a long-acting form of alpha interferon) plus ribavirin in treating hepatitis C (genotype 1) infection with and without kidney disease.

DETAILED DESCRIPTION:
Up to 105 patients with chronic hepatitis C will be enrolled in a study of the combination of pegylated alpha interferon and ribavirin for 48 weeks with the option of early discontinuation of therapy for patients who do not respond within 24 weeks of starting therapy. Adult patients will be chosen who have chronic hepatitis C, HCV RNA in serum, HCV genotype 1 and liver histology showing chronic hepatitis C. Patients with advanced liver disease and clinical decompensation and patients who have received alpha interferon in the past will not be eligible. The 100 patients will consist of four groups: Groups A, B and D will comprise 25 patients each with typical uncomplicated chronic hepatitis C; Group C will comprise 25 patients with renal insufficiency or renal failure on chronic dialysis awaiting kidney transplantation. Group D will comprise up to 30 patients with typical uncomplicated chronic hepatitis C. After medical evaluation and liver biopsy, patients will begin receiving pegylated alpha interferon (peginterferon) by subcutaneous injection in a dose of 180 mcg per week. After the initial injection, patients will have blood taken and symptoms recorded at 12, 24, 48, 72 hours and weekly thereafter for four weeks. Patients in Groups A, B and C will receive peginterferon weekly, whereas patients in Group D will receive it twice weekly in a reduced dose (90 mcg per injection) for the first 4 weeks of treatment and weekly in a dose of 180 mcg per injection thereafter. Patients in Groups A and D will also begin receiving ribavirin orally in a dose of 1000 mg (if body weight is less than 75 kg) or 1200 mg daily (if body weight greater than or equal to 75 kg) given in capsules of 200 mg twice daily starting with the first dose of peginterferon. Patients in Group B will start ribavirin in the doses given above after the first month of therapy (with the fifth injection: week 4). Patients in Group C (renal disease) will start ribavirin in a dose of 200 mg daily after the first month (week 4) of therapy; in this group the dose of ribavirin will be gradually increased at 4 week intervals on the basis of tolerance (hemolysis and anemia). During the initial 24-week period of combination therapy, patients will be seen in the outpatient clinic for medical interview, physical examinations and blood tests at 2 to 4 week intervals. At 24 weeks, patients will be classified as either responders or non-responders based upon HCV RNA testing. Both groups will be offered therapy for another 24 weeks (total treatment = 48 weeks). Because sustained responses are rare in patients who have not become HCV RNA negative by 24 weeks, non-responders will be offered the option of stopping therapy early and being followed on no therapy. After stopping therapy, patients will be followed at 1 to 2 month intervals and undergo repeat medical evaluation (without liver biopsy) at the 72 week point (18 months after enrollment).

The primary criterion for success of therapy overall will be sustained loss of HCV RNA as assessed at 18 months. Secondary criteria will be normalization of ALT levels and improvement of symptoms. This study will allow for therapy of patients with chronic hepatitis C with the combination of peginterferon and ribavirin demonstrating whether early viral kinetics are predictive of outcome of therapy. This study will also allow for comparison of the kinetics of loss of HCV RNA comparing peginterferon alone to peginterferon with ribavirin, peginterferon given once weekly to peginterferon given twice weekly, and comparing kinetics between patients with and without renal disease. The study will also allow for assessment of the safety of addition of ribavirin in patients with renal compromise.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Patients:

* Age 18 years or above, male or female.
* Presence of HCV RNA (with or without anti-HCV) in serum.
* Genotype 1 HCV as determined by probe specific hybridization (Inno-Lipa assay).
* Evidence of chronic hepatitis on liver biopsy done within the previous 48 months with a necroinflammatory histology activity index of at least 3 (out of a maximum of 18).
* Written informed consent.

Additional inclusion criteria for Groups A, B and D:

- Serum alanine (ALT) or aspartate aminotransferase (AST) above the upper limit of the normal range (ALT 41 greater than IU/L: AST greater than 31 IU/L) on any serum testing during the previous six months.

Additional inclusion criteria for Group C:

* Chronic renal disease with creatinine clearance less than 50 cc/min or serum creatinine greater than 2.0 mg%.
* If on chronic hemodialysis or peritoneal dialysis, stable clinical condition including stable hematocrit.
* If on chronic dialysis, potential candidacy for renal transplantation.

EXCLUSION CRITERIA:

* Previous treatment with alpha interferon.
* If cirrhosis is present, decompensated liver disease, as marked by bilirubin greater than 4 mg%, albumin less than 3.0 gm%, prothrombin time greater than 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy.
* Serum ALT or AST levels greater than 1000 U/L (greater than 25 times ULN). Such patients will not be enrolled but may be followed until three determinations are below this level.
* Pregnancy or, in women of child-bearing potential or in spouses of such women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicide, or birth control pills, or an intrauterine device.
* Significant systemic or major illnesses other than renal failure (in Group C), including congestive heart failure, organ transplantation, serious psychiatric disease or depression, human immunodeficiency virus (HIV) infection, and angina pectoris.
* Pre-existing anemia (hematocrit less than 33%) or known history of hemolytic anemia. In patients in Group C, erythropoetin therapy will be modified to achieve an adequate hematocrit if clinically indicated.
* Other antiviral therapy within the last 6 months.
* Immunosuppressive therapy with either corticosteroids (more than 5 mg of prednisone daily) or major immunosuppressive agents (such as azathioprine or 6-mercaptopurine).
* Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, Wilson's disease, alcoholic liver disease, hemochromatosis, alpha-1-antitrypsin deficiency).
* Evidence of coronary artery disease or cerebral vascular disease, including abnormalities on exercise stress testing in patients with defined risk factors who will be screened for evidence of underlying coronary artery disease.
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.
* Evidence of hepatocellular carcinoma; either alphafetoprotein (AFP) levels greater than 50 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.
* Clinical gout.
* Active, serious autoimmune disease such as lupus erythematosis, ulcerative colitis, Crohn's disease or rheumatoid arthritis that in the opinion of the investigators might be exacerbated by therapy with alpha interferon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, MD, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Liang TJ, Rehermann B, Seeff LB, Hoofnagle JH. Pathogenesis, natural history, treatment, and prevention of hepatitis C. Ann Intern Med. 2000 Feb 15;132(4):296-305. doi: 10.7326/0003-4819-132-4-200002150-00008. PMID 10681285
- [Background] Major ME, Feinstone SM. The molecular virology of hepatitis C. Hepatology. 1997 Jun;25(6):1527-38. doi: 10.1002/hep.510250637. No abstract available. PMID 9185778
- [Background] Kiyosawa K, Sodeyama T, Tanaka E, Gibo Y, Yoshizawa K, Nakano Y, Furuta S, Akahane Y, Nishioka K, Purcell RH, et al. Interrelationship of blood transfusion, non-A, non-B hepatitis and hepatocellular carcinoma: analysis by detection of antibody to hepatitis C virus. Hepatology. 1990 Oct;12(4 Pt 1):671-5. doi: 10.1002/hep.1840120409. PMID 2170265
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-DK-0065.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon+Ribavirin: peginterferon alpha-2a, 180 ug subcutaneous once weekly and weight-based oral ribavirin (1000 mg daily for patients less than 75 kg and 1200 mg daily for patients greater than 75 kg) for 48 weeks
- Peginterferon Alone: peginterferon-alpha 2a, 180 ug subcutaneous once weekly for the first 4 weeks of therapy, after which peginterferon was continued at the same dose and weight-based oral ribavirin was added and continued for an additional 44 weeks.
Period: Overall Study
Arm/Group | Peginterferon+Ribavirin | Peginterferon Alone
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon+Ribavirin | Peginterferon Alone | Total
Number analyzed (Participants) | 25 | 25 | 50
Age Continuous [Median (Full Range); unit: years] | 49 [35 to 68] | 52 [28 to 67] | 51 [28 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 14 | 10 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 17 | 21 | 38
  African American | 4 | 2 | 6
  Asian | 2 | 1 | 3
  Hispanic | 2 | 1 | 3
Duration of infection [Mean (Standard Deviation); unit: year] | 23 (9.0) | 23 (7.7) | 23 (8.4)
Mode of infection [Number; unit: participants]
  Injection drug use | 10 | 8 | 18
  Blood transfusion | 8 | 9 | 17
  Other | 5 | 6 | 11
  Unknown | 2 | 2 | 4
Weight [Mean (Standard Deviation); unit: kg] | 78.1 (17) | 76.8 (19) | 77.5 (18.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/(m^2)] | 26.9 (4.9) | 27.0 (4.8) | 27.0 (4.9)
Alanine transaminase [Mean (Standard Deviation); unit: U/L] | 69 (61) | 96 (79) | 83 (71)
Ishak fibrosis [Number; unit: participant] — Fibrosis was staged with the Ishak scale (ranging from 0 = no fibrosis to 6 = cirrhosis). Higher values represent a worse outcome.
  participant
    0-2 | 15 | 16 | 31
    3-6 | 10 | 9 | 19
Histology activity index [Median (Full Range); unit: Units on a scale] — Possible range 0-18. Higher values represent a worse outcome.
  Units on a scale | 8 [5 to 13] | 8 [3 to 15] | 8 [3 to 15]
Hepatitis C Virus RNA level [Mean (Standard Deviation); unit: log(IU/mL)] | 6.2 (0.53) | 6.2 (0.58) | 6.2 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatitis C Virus RNA Levels During Phase I
Time Frame: From day 0 to day 3
Measure: Median (Full Range); unit: log(IU/mL)
Arm/Group | Peginterferon+Ribavirin | Peginterferon
Number analyzed (Participants) | 24 | 24
log(IU/mL) | 0.50 [-0.40 to 2.30] | 0.70 [-0.10 to 1.70]
Statistical Analysis 1: Comparison: Peginterferon+Ribavirin vs Peginterferon; Null hypothesis: there is no difference in the outcome between the two groups; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Peginterferon+Ribavirin | Peginterferon Alone
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes